CLINICAL TRIAL: NCT03178539
Title: Comparative Study Between the Effect of Diclofanic and Ketorolac in Post Tonsillectomy Pain Management
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, assistant professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17100114
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Pain, Acute
Keywords: tonsillectomy; post operative analgesia; diklofanic; ketorolac
MeSH Terms: conditions — Acute Pain | interventions — Diclofenac; Ketorolac; Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- diclofenac (Active Comparator): patients will receive intra-operative diclofenac sodium at dose of 0.3 mg/kg intravenously then will continue postoperatively on the same drug received intra-operative.
  Interventions: Drug: diclofenac
- ketorolac (Active Comparator): patients will receive intra-operative ketorolac tromethamine at dose of 0.5 mg/kg intravenously then will continue postoperatively on the same drug received intra-operative.
  Interventions: Drug: ketorolac

INTERVENTIONS:
Drug: diclofenac — non steroidal anti-inflammatory drug
  Other Names: Voltaren
  Arms: diclofenac
Drug: ketorolac — non steroidal anti-inflammatory drug
  Other Names: Tromethamine
  Arms: ketorolac

SUMMARY:
Compare between the analgesic efficacy of diclofenac sodium and ketorolac tromethamine in post-tonsillectomy pain management.and Compare between the effect of diclofenac sodium and ketorolac tromethamine on post-tonsillectomy bleeding

DETAILED DESCRIPTION:
patients will be randomly allocated to two groups of 50 patients each Group (A): will receive intra-operative diclofenac sodium at dose of 0.3 mg/kg intravenously.

Group (B): will receive intra-operative ketorolac tromethamine at dose of 0.5 mg/kg intravenously.

Then the two groups will continue postoperatively on the same drug received intra-operative

I. Intra-operative data:

Bleeding score will be assessed by the surgeon at the end of the operation using the following Scale for bleeding assessment (0 = no bleeding, 1 = bleeding as usual, 2 = bleeding more than usual, 3 = profuse, 4 = excessive, and lastly 5 = excessive and continuous).

II. Early Post-operative data:

1. Post- tonsillectomy bleeding assessments;

   * Bleeding score will be recorded immediately postoperative and 3, 6, 12 and 24h postoperatively.
   * Hospital re-admission because of bleeding.
   * Re-operation because of bleeding.
2. Post- tonsillectomy pain assessments; Pain intensity will be assessed postoperatively by the verbal rating scale (VRS; 0 = no pain, 1 = mild pain, 2 = moderate pain, 3= severe pain, and lastly 4= excruciating pain). VRS assessment will be performed immediately postoperative and 3, 6, 12 and 24h postoperatively. Analgesia will be given if requested or if the VRS≥3. Patients in Group A will receive diclofenac sodium 0.3 mg/kg iv, while patients in Group B will receive ketorolac tromethamine 0.5 mg/kg.

The total consumption of analgesics used in each group in the first 24 h postoperative will be calculated and the time of the first request for analgesia will be recorded.

- Time needed to restore normal dietary habits.

IV. Late Post-operative data:

As aweekly follow up for 2 weeks :

1. bleeding tendency
2. Dysphagia.

   * Time needed to restore normal dietary habits

ELIGIBILITY:
Inclusion Criteria:

* Children scheduled for elective tonsillectomy\adenotnsillectomy for chronic or recurrent tonsillitis and aged between 6 to 12 years

Exclusion Criteria:

* Known hypersensitivity to medication drugs.
* Coagulation disorders, thrombocytopenia or active bleeding for any cause.
* Bronchial asthma.
* Significant cardiac, renal, pulmonary, hepatic disease or peptic ulcer.
* The use of any analgesic medications within 24h preoperative or antiplatelet medication within the past 2 weeks.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
pain relieve | 24 hours
  the verbal rating scale (VRS; 0 = no pain, 1 = mild pain, 2 = moderate pain, 3= severe pain, and lastly 4= excruciating pain). VRS assessment will be performed immediately postoperative and 3, 6, 12 and 24h postoperatively

SECONDARY OUTCOMES:
bleeding | two weeks
  Bleeding score will be assessed by the surgeon at the end of the operation using the following Scale for bleeding assessment (0 = no bleeding, 1 = bleeding as usual, 2 = bleeding more than usual, 3 = profuse, 4 = excessive, and lastly 5 = excessive and continuous).
dysphagia | two weeks
  time needed to restore normal dietary habbit

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel_Ghaffar, MD, Principal Investigator — Assistant professor, faculty of medicine, Assiut university
Locations (1):
- Assiut university hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No